CLINICAL TRIAL: NCT07257055
Title: Phase 2 Study of BTKi-Rituximab Induction Followed by Glofitamab Consolidation in High Risk Untreated MCL Patients - WINDOW-4 Study
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-0423; NCI-2025-08762 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2025-11-21; First posted 2025-12-02 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Phase 2 Study; MCL; BTKi; Rituximab; Glofitamab
MeSH Terms: interventions — acalabrutinib; zanubrutinib; Rituximab; glofitamab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- 1-Induction (Experimental): Phase 2 Induction Treatment with BTKi-R - Rituximab/Ruxience + Acalabrutinib/Zanubrutinib
  Interventions: Drug: Acalabrutinib; Drug: Rituximab
- 2-Consolidation (Experimental): Phase 2 Consolidation Treatment with Glofitamab
  Interventions: Drug: Glofitamab
- 3-Maintenance (Experimental): Phase 2 Maintenance Treatment with BTKi-R - Rituximab/Ruxience + Acalabrutinib/Zanubrutinib
  Interventions: Drug: Acalabrutinib; Drug: Rituximab

INTERVENTIONS:
Drug: Acalabrutinib — Given by po
  Other Names: Zanubrutinib
  Arms: 1-Induction; 3-Maintenance
Drug: Rituximab — Given by IV
  Other Names: Ruxience
  Arms: 1-Induction; 3-Maintenance
Drug: Glofitamab — Given by IV
  Arms: 2-Consolidation

SUMMARY:
to learn if giving glofitamab after treatment with BTKi-rituximab can help to control high-risk MCL.

DETAILED DESCRIPTION:
Primary Objective To determine the rate of minimal residual disease (MRD) negativity following treatment with 12 cycles of glofitamab in participants with high risk MCL after achieving CR on standard first line treatment with BTKi (Acalabrutinib or Zanubrutinib)-rituximab

Secondary Objectives To determine overall response rate (ORR), complete response (CR), Early MRD negative response, progression-free survival (PFS), overall survival (OS), and evaluate the safety of glofitamab as consolidation treatment for MCL

ELIGIBILITY:
Eligibility Criteria

Participants must meet the following criteria for study entry:

1. Confirmed diagnosis of mantle cell lymphoma by hematopathology. MCL should have CD20 positivity (by flow or IHC in tissue or in BM) with presence of chromosome translocation t (11;14), (q13;q32) and/or overexpression of cyclin D1 in tissue biopsy. Cyclin D negative MCL are allowed after discussion with study PI.
2. Participants should have a life expectancy >= 12 weeks.
3. Newly diagnosed, untreated, high risk participant without any prior therapy for MCL and are eligible to receive BTKi-R and glofitamab therapy.
4. High risk MCL (Blastoid/pleomorphic histology, high Ki-67 (≥50%), TP53/NOTCH1/2, NSD2, UBR5, TRAF2, SP140, SMARCA4, KMT2D, BIRC3 mutated or any of these mutations or more than 2 mutations with some evidence of prognostic impact, complex karyotype and/or Bulky nodal disease >= 5 cm or spleen >= 20 cm, FISH positive for TP53 or MYC from involved tissues or TP53 and MYC positive intensity in lymphoma cells in involved tissues (positive by hem-path criteria at MDACC), high risk MIPI score (with/without Ki-67%). Presence of any or all of these features would qualify as high risk but will need to be reviewed and approved by the study PI.

6. Participants who are willing and able to participate in all required evaluations and procedures in this study protocol, including swallowing capsules and tablets without difficulty.

7. Understand and voluntarily sign an IRB-approved informed consent form. 8. Age ≥ 18 years at the time of signing the informed consent. 9. Bi-dimensional measurable disease using the 2014 Cheson criteria (Measurable disease by PETCT scan or CT scan (if PET-CT not approved and study PI approves) defined as at least 1 lesion that measures ≥ 1.5 cm in single dimension.) and/or spleen only involved (>=20 cm). Leukemic phase MCL are allowed without bulky measurable disease if they have other high-risk features after discussion with the study PI. These participants are allowed if they meet any other high-risk features, determined by the study PI.

10. Eastern Cooperative Oncology Group (ECOG) performance status of 1 or less. 11. Participants with preexisting well-controlled cardio-vascular comorbidities - participants on anticoagulants (excluding warfarin and vitamin K antagonists), antiplatelet, antihypertensive, prior ablation, anti-arrhythmia, prior arrhythmias, baseline EKG abnormalities and cardiology clearance are allowed. Ejection fraction >=50% and cardiology evaluation is needed. (Echo and EKG and cardiology consultation within 2 months prior to C1D1 are allowed).

12. An absolute neutrophil count (ANC) > 1,000/mm3 and platelet count >100,000/mm3 (Participants who have >50% bone marrow or spleen infiltration by MCL are eligible if their ANC is ≥ 500/mm3 [growth factor allowed] or their platelet level is equal to or >= than 30,000/mm3 (transfusions allowed) These participants should be discussed with the PI of the study for final approval). Hemoglobin > 8.0 g/dL (> 80 g/L), unsupported for 2 days before first treatment (unless attributable to the underlying disease as determined by the study PI) 13. Serum bilirubin <1.5 mg/dl, AST (SGOT) and ALT (SGPT) < 2.5 x upper limit of normal or < 5 x upper limit of normal if hepatic metastases are present. Gilbert's disease is allowed.

14. Creatinine clearance. >=30 mL/min (by 2021 chronic kidney disease epidemiology (CKD-EPI) creatinine equation or 2021 CKD-EPI creatinine-cystatin C equation., APPENDIX VI I) 15. Contraception in female participants of childbearing potential- female participants must remain abstinent or use contraceptive methods with a failure rate of < 1% per year during the treatment period and for at least 6 months after pretreatment with obinutuzumab, 2 months after the final dose of glofitamab and 2 months after the final dose of tocilizumab (as applicable), whichever is longer. Women must refrain from donating eggs during this same period.

16. A female participant is considered to be of childbearing potential if she is postmenarchal, has not reached a postmenopausal state (³ 12 continuous months of amenorrhea with no identified cause other than menopause), and is not permanently infertile due to surgery (i.e., removal of ovaries, fallopian tubes, and/or uterus) or another cause as determined by the investigator (e.g., Müllerian agenesis). Per this definition, a female participant with tubal ligation is considered to be of childbearing potential. The definition of childbearing potential may be adapted for alignment with local guidelines or regulations.

17. Examples of contraceptive methods with a failure rate of < 1% per year include bilateral tubal ligation in female of child-bearing potential, male sterilization, hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices.

18. Hormonal contraceptive methods are also recommended to be supplemented by a barrier method.

19. The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the individual. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not adequate methods of contraception. If required per local guidelines or regulations, locally recognized adequate methods of contraception and information about the reliability of abstinence will be described in the local Informed Consent Form.

20. Contraception for male participants: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods, and agree to refrain from donating sperm, as defined below: 21. With a female partner of childbearing potential or pregnant female partners, male participants must remain abstinent or use a condom plus an additional contraceptive method that together result in a failure rate of < 1% per year during the treatment period and for at least 6 months after pretreatment with obinutuzumab, 2 months after the final dose of glofitamab or 2 months after the last dose of tocilizumab (as applicable), whichever is longer. Male participants must refrain from donating sperm during this same period.

22. The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the individual. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not adequate methods of contraception. If required per local guidelines or regulations, locally recognized adequate methods of contraception and information about the reliability of abstinence will be described in the local Informed Consent Form. ..

a. Females must agree to abstain from breastfeeding during study participation and for at least 12 months after glofitamab discontinuation. Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test. WOCBP and males must be willing to use highly effective methods of birth control. Woman of childbearing potential (WOCBP) who are sexually active must use highly effective methods of contraception during treatment and 1 week after the last dose of acalabrutinib b. Females of childbearing potential (FCBP§ ) must: i. Have one negative pregnancy tests via serum in some cases urine (as clinically indicated) one week or immediately prior to starting study therapy. She must agree to ongoing pregnancy testing during the course of the study, prior to day 1 of each cycle, and after end of study therapy. This applies even if the subject practices true abstinence* from heterosexual contact.

ii. Not engaging in sexual activity for the total duration of the trial and the drug washout period is an acceptable practice. Otherwise, she must agree to use, and be able to comply with highly effective contraception.

c. Male subjects must: i. A male subject who is sexually active with a female with reproductive potential is also recommended to use a barrier method of birth control, eg, either condom with spermicidal foam/gel/film/cream/suppository or partner with occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/ suppository (including dose interruptions), even if they have undergone a successful vasectomy, from the time of signing consent and for at least 2 months after the last dose of glofitamab, 6 months after treatment with obinutuzumab, or 2 months after the last dose of tocilizumab (if applicable), whichever is longer. For male participants with a pregnant or non-pregnant WOCBP partner, should use barrier contraception, during treatment and for 1 week after the last dose of acalabrutinib, 180 days following the last dose of rituximab, 2 months following the last dose of glofitamab,6 months following the last dose of obinutuzumab, 2 months following the last dose of tocilizumab (if applicable), , whichever is longer, even if they have had a successful vasectomy.) d. Participant must be willing and able to comply with protocol-mandated hospitalization upon administration of the first dose of glofitamab. e. f. Have achieved complete metabolic response by Lugano criteria[35] to go to part 2 for glofitamab consolidation g. Performance status ≤1 on the ECOG scale h. All subjects must i. Agree to refrain from donating blood while on study treatment, during dose interruptions and for at least 12 months following the last dose of study treatment.

Exclusion Criteria Having radiologically confirmed relapsed/refractory disease.

1. Isolated bone marrow or GI only disease MCL participants and/or lack of any measurable disease, except if participants have leukemic phase MCL with any high risk features.
2. Pregnant or breast-feeding females.
3. Participants who are primary refractory to BTKi-R (No response/progressive disease within first 3 months of BTKi-R)
4. Received any investigational drug within 30 days or 5 half-lives (whichever is shorter) before first dose of study drug.
5. Current life-threatening illness, medical condition, or organ system dysfunction which, in the Investigator's opinion, could compromise the subject's safety or put the study at risk.
6. Known HIV infection.
7. Known history of hemophagocytic lymphohistiocytosis (HLH)
8. Known or suspected chronic active Epstein-Barr virus infection (clearance with infectious disease is needed to allow these participants)
9. Positive SARS-CoV-2 test within 7 days prior to enrollment. Rapid antigen test result is also acceptable.
10. Participants who do not meet high risk features as indicated above in inclusion.
11. Hepatitis B or C serologic status: subjects who are hepatitis B core antibody (anti-HBc) positive and who are hepatitis B surface antigen (HBsAg) negative will need to have a negative polymerase chain reaction (PCR) and must be willing to undergo DNA PCR testing during the study to be eligible. Those who are HBsAg positive or hepatitis B PCR positive will be excluded (unless cleared by hepatology and ID team after discussion with study PI). Subjects who are hepatitis C antibody positive will need to have a negative PCR result to be eligible. Those who are hepatitis C PCR positive will be excluded.
12. Prior malignancy (or any other malignancy requiring active treatment), except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, in situ ca prostate, in situ melanoma (> 5 mm margins) or other cancer from which the subject has been disease free for ≥ 3 years or which will not limit survival to < 3 years or not on active systemic chemotherapy.
13. Central nervous system involvement with mantle cell lymphoma or with suspected or confirmed progressive multifocal leukoencephalopathy (PML). Magnetic resonance imaging (MRI) of the brain, if performed, showing evidence of central nervous system (CNS) lymphoma or Lumbar puncture with flow cytometry, if performed, with CSF involvement.
14. History or presence of uncontrolled CNS disorder, such as seizure disorder, cerebrovascular ischemia/hemorrhage, dementia, cerebellar disease, cerebral edema, posterior reversible encephalopathy syndrome, or any autoimmune disease with CNS involvement.
15. Active bleeding, history of bleeding diathesis (such as Hemophilia or Von-Willebrand disease), Any history of intracranial bleed or stroke within 6 months of first dose of study drug.
16. Uncontrolled AIHA (autoimmune hemolytic anemia) or ITP (idiopathic thrombocytopenic purpura).
17. Malabsorption syndrome, disease which is clinically significantly affecting gastrointestinal function, or resection of the stomach or small bowel or active ulcerative colitis, symptomatic inflammatory bowel disease, or partial or complete bowel obstruction, or any other gastrointestinal condition that could interfere with the absorption and metabolism of BTKi. These participants may be allowed after discussion, clearance with GI team and discussion with the study PI.
18. Presence of a clinically significant gastrointestinal ulcer diagnosed by endoscopy within 3 months before first dose of study drug.
19. Requires anticoagulation with warfarin or equivalent vitamin K antagonist, active treatment for pulmonary embolism (PE)/ deep vein thrombosis (DVT) and persons with mechanical cardiac valves. These participants may be allowed after review with benign hematology and study PI.
20. Concomitant use of corticosteroids at > 20 mg prednisone or equivalent per day longer than 2 weeks.
21. Primary immunodeficiency which is clinically active
22. History of confirmed autoimmune disease (e.g. Crohn's disease, rheumatoid arthritis, systemic lupus) resulting in end organ injury or requiring systemic immunosuppression/systemic disease modifying agents within the last 2 years. Rheumatology clearance and approval by study PI is required for pts with remote history of auto-immune disease.
23. The use of strong CYP3A inhibitors within 1 week or strong CYP3A inducers within 3 weeks of the first dose of study drug is prohibited.
24. Requires treatment with strong CYP3A inhibitors or inducers.
25. Clinically significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of Screening, or any Class 3 (moderate) or Class 4 (severe) cardiac disease as defined by the New York Heart Association (NYHA) Functional Classification. Subjects with controlled, asymptomatic heart failure during screening can enroll on study and/or any of the following cardiac related conditions, unless cleared by cardiology and study PI:
26. NYHA Class III and IV heart failure,
27. Active/symptomatic coronary artery disease,
28. Myocardial infarction in the preceding 6 months,
29. Significant conduction abnormalities, including but not limited to:
30. Left bundle branch block,
31. 2nd degree AV block type II,
32. 3rd degree block,
33. QT prolongation (QTc > 500 msec),
34. Sick sinus syndrome,
35. Ventricular tachycardia,
36. Symptomatic bradycardia (heart rate < 50 bpm),
37. Persistent and uncontrolled atrial fibrillation.
38. Uncontrolled hypertension
39. Uncontrolled Hypotension
40. Light headedness and syncope,
41. Acute infection requiring systemic anti-infective treatment systemic antibiotics, antivirals, or antifungals, or including subjects with positive cytomegalovirus [CMV] DNA polymerase chain reaction [PCR] within 14 days prior to initiation of therapy. Participant who exhibit active uncontrolled infection on BTKi-R alone will not be excluded but would await adequate infection control and then get CAR T, as long as they have evidence of disease.
42. Vaccinated with live, attenuated vaccines within 6 weeks of first dose of study drug.
43. Any other serious medical condition including, but not limited to, clinically significant uncontrolled diabetes mellitus, COPD, renal failure, psychiatric illness or social circumstances that, in the investigator's opinion places the participant at unacceptable risk and would prevent the participant from signing the informed consent form or complying with study procedures.
44. Known history of hypersensitivity or anaphylaxis to study drug(s) including active product or excipient components.

6. Concurrent participation in another therapeutic clinical trial. 47. Is unable to swallow any oral medication or has clinically significant gastrointestinal disease thatwould limit absorption of oral medication.

48. . 49. Major surgical procedure within 28 days of first dose of study drug. Note: If a subject had major surgery, they must have recovered adequately from any toxicity and/or complications from the intervention before the first dose of study drug.

50. Participants with inactive hepatitis B infection must adhere to hepatitis B reactivation prophylaxis unless contraindicated. Hepatitis B or C serologic status: subjects who are hepatitis B core antibody (antiHBc) positive and who are surface antigen negative will need to have a negative polymerase chain reaction (PCR). Those who are hepatitis B surface antigen (HbsAg) positive or hepatitis B PCR positive will be excluded. Subjects who are hepatitis C antibody positive will need to have a negative PCR result. Those who are hepatitis C PCR positive will be excluded. Subjects with a history of Hepatitis C who received antiviral treatment are eligible as long as PCR is negative.

1. History of severe allergic or anaphylactic reactions or intolerance to anti-CD20 monoclonal antibody therapy or any bispecific antibody.
2. History of immunodeficiency (except for hypogammaglobulinemia) or concurrent systemic immunosuppressant therapy (e.g., cyclosporine, tacrolimus, etc., or chronic administration glucocorticoid equivalent of >10mg/day of prednisone) within 28 days of the first dose of study drug with exception of steroid used for IV contrast allergy. In addition, use of inhaled, topical, intranasal corticosteroids or local steroid injection (eg, intra- articular injection) is permitted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-05-12 (Estimated); Primary Completion 2028-11-24 (Estimated); Study Completion 2030-11-24 (Estimated)

PRIMARY OUTCOMES:
Safety and adverse events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Preetesh Jain, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org